CLINICAL TRIAL: NCT05512858
Title: Exploring the Effectiveness of a Sensory Room in Reducing Seclusion, Restraint and Aggression at an Acute Psychiatric Unit
Brief Title: Sensory Room at an Acute Psychiatric Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Aviv University (Other)
Collaborators: Abarbanel Mental Health Center (Other Government)
Responsible Party: Principal Investigator, Tami Bar-Shalita, Principal Investigator, Tel Aviv University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 164
Record Dates: First submitted 2022-07-25; First posted 2022-08-23 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Psychiatric Disorder
Keywords: psychiatric disorder; sensory processing; sensory room; seclusion; restraint; aggression; acute psychiatric ward
MeSH Terms: conditions — Mental Disorders; Aggression

STUDY DESIGN:
Intervention Model Description: Two phases, First with no intervention (=control group), second with intervention(study group).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- phase 1 (No Intervention): Data on restrictions and aggression events in the department will be collected throughout the two phases, and the participants will undergo an evaluation process.
- phase 2 (Experimental): Data on restrictions and aggression events in the department will be collected throughout the two phases, and the participants will undergo an evaluation process. n addition, the subjects who participate in the intervention will wear an Empatica-E4 wristband to monitor autonomous metrics during their stay in the sensory stimulation room and will undergo a brief interview regarding their experience using the room.
  Interventions: Behavioral: sensory room

INTERVENTIONS:
Behavioral: sensory room — the room has dimmed lighting, sensing games, essential oils, picture books and cookbooks, two heavy blankets (weighing 9 kg and 11 kg), a rocking chair, and a vestibular plate. The occupational therapist will accompany the first entry into the room to create a sensory profile, adjust and instruct on the means, and write a treatment card. The treatment card will record the patient's choices and instructions for arranging the room, and it will be used by the staff members who will admit the patient as needed. Each patient will be able to stay in the room for self-treatment according to the individual treatment card prepared at the first sensory room treatment, up to half an hour.
  Arms: phase 2

SUMMARY:
the aim of the presented study is to explore the effectiveness of a sensory room in reducing seclusion, restraint and aggression at an acute psychiatric ward.

DETAILED DESCRIPTION:
Background In recent years, there has been an increase in violence in mental health centers in Israel. Until recently, the phenomenon was treated under mechanical restrictions and patient isolation. Today the trend is to reduce the use of restrictions, with the main alternative being the provision of medication and de-escalation techniques, one of which is sensory stimulation using sensory rooms. A sensory room in the psychiatric unit has been found as an effective intervention for reducing patients' distress and aggression. However, the effectiveness of using the room has not yet been studied in Israel and in relation to pain.

Method

The experimental study will be conducted in two phases each lasting three months in an acute psychiatric ward:

1. Without intervention (control group).
2. With intervention. Data on restrictions and aggression events will be collected throughout the two phases, and the participants will undergo an evaluation process using self reports.

In addition,subjects who will participate in the intervention (study group) will wear an Empatica-E4 wristband to monitor autonomous metrics during their stay in the sensory stimulation room and will undergo a brief interview regarding their experience using the room.Thus the intervention phase (Study group) will comprise mixed methods.

Population Eighty men aged 18-50, a convenience sample, who speaks Hebrew; treated with psychiatric medication for at least two weeks; and hospitalized for up to 70 days.

Expected results:

Statistical significant group differences will be found in the sum of ward restrictions (i.e., sedatives, physical restraint, and seclusion), showing less during phase 2 (study group): The study group (2nd phase) will receive fewer sedatives and use less physical restraint and seclusion.

Statistical significant group differences will be found in the aggression incidents showing fewer reports of aggression in the study group.

Statistical significant differences will be found in the HRV indices between pre and post sensory room treatment, showing reduced values post treatment.

statistically significant correlations will be found between sensory over-responsivity and the number of aggression events so that higher sensory responsiveness (SOR) will be correlated with more aggression events.

statistically significant correlations will be found between sensitivity to pain and the number of aggression incidents: higher pain sensitivity will be correlated with fewer incidents of aggression.

ELIGIBILITY:
Inclusion Criteria:

* Hebrew language Proficiency receiving psychiatric medication of any kind regularly for at least 14 days hospitalized in full hospitalization for up to 70 days.

Exclusion Criteria:

* chronic pain, neurodevelopmental syndrome active use of psychoactive substances.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2022-08-28 (Actual); Primary Completion 2023-06-25 (Actual); Study Completion 2023-06-25 (Actual)

PRIMARY OUTCOMES:
Number of restrictions | through study completion, an average of 1 year
  In this study, restrictions are defined as incidents of entering confinement in an isolation room and as taking additional sedative medication. The data collection for the entrance to isolation and tying rooms will be done through a tying notebook managed by the nursing staff; in the notebook, the events are recorded and signed by a doctor. Monitoring of taking the additional drug treatment will be done through the center's computerized system.
Number of aggression events | through study completion, an average of 1 year
  Aggression incidents are "exceptional incidents" in the ward, an incident in which a person or an object was harmed. These events are logged in the center's computer system.

SECONDARY OUTCOMES:
Interview - qualitative measure | after every intervention, an average of six months
  In order to understand the subject's experience of using the room, an occupational therapist will conduct a semi-structured five-question interview when the subject leaves the sensory stimulation room.
Emptica-E4- physiological parameter (EDM) | during the intervention, an average of six months
  A medical-grade wearable device that offers real-time physiological data acquisition. Wearable tool, bracelet, battery chargedwill be used to measure electrodermal activity (EDM). Data will automatically be uploaded to E4 connect, a cloud platform after the session ends. The analysis will be done using Kubios software.
Emptica-E4- physiological parameter (PPG) | during the intervention, an average of six months
  A medical-grade wearable device that offers real-time physiological data acquisition. Wearable tool, bracelet, battery charged, will be used to measure Blood Volume Pulse (BVP), from which heart rate variability can be derived. Data will automatically be uploaded to E4 connect, a cloud platform after the session ends. The analysis will be done using Kubios software.

OTHER OUTCOMES:
Clinical Global Impression (CGI) | through study completion, an average of 1 year. Will be filled out for each participant once
  A reliable and valid standard evaluation designed to assess the severity of psychiatric illness. The tool consists of three items: CGI-Severity of Illness (CGI-S), CGI-Global Improvement, and CGI-Efficacy Index ; only CGI-S will be used in this study. The psychiatrist should indicate in the range between 1 ("normal, no evidence of disease") and 7 ("among the most severe cases of patients") the patient's condition compared to patients with the same diagnosis with regards to the following parameters: symptoms, behavior, and function in the last week.
Montreal Cognitive Assessment (MoCA) | through study completion, an average of 1 year. Each participant will answer once
  A 10-minute cognitive screening tool assessment for detecting cognitive impairment. The MoCA items include short term memory recall, visuospatial ability, executive function, attention-concentration-working memory, language, and orientation to time and place.
The Sensory Responsiveness Questionnaire Intensity Scale (SRQ-IS) | through study completion, an average of 1 year. Each participant will answer once
  A 58-item questionnaire aimed at clinically classifying sensory modulation dysfunction in adults. Items represent typical daily life situations involving auditory, visual, gustatory, olfactory, vestibular and somatosensory sensations, excluding pain. Items are phrased either in a hedonic or aversive valence and are graded on a 5-point Likert scale: 'not at all' (1) to 'very much' (5). Two cut-off scores are provided.
Pain Sensitivity Questionnaire (PSQ) | through study completion, an average of 1 year. Each participant will answer once
  A 17 item questionnaire aimed to quantify everyday somatosensory pain sensitivity to imagined painful daily life situations. Participants rate the intensity of imagined pain on a 10-point scale: 'not painful at all' (0) to 'the worst pain imaginable' (10). The Pain Sensitivity Questionnaire provides a total score and two sub-scores.
State-Trait Anxiety Inventory (STAI) | through study completion, an average of 1 year. Each participant will answer once
  Self-report questionnaire designed to determine the anxiety level of a patient and divides anxiety into state and trait anxieties. This study will use STAI-T only. Trait anxiety is the presence of disproportionately long-term and severe anxiety related to an objective cause. STAI has 20 items, each item is rated on a scale of 1 to 4, and the sum of all items determines the anxiety level. A score in the range of 20-80 is considered a high score and indicates intense anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Liron Peretz, BOT, Study Chair — Tel Aviv University
Locations (1):
- Abarbanel Mental Health Center, Bat Yam, Israel

IPD SHARING:
Plan to Share IPD: No
Data will be available upon personal request

REFERENCES:
- [Background] Barton SA, Johnson MR, Price LV. Achieving restraint-free on an inpatient behavioral health unit. J Psychosoc Nurs Ment Health Serv. 2009 Jan;47(1):34-40. doi: 10.3928/02793695-20090101-01. PMID 19227108
- [Background] Berk M, Ng F, Dodd S, Callaly T, Campbell S, Bernardo M, Trauer T. The validity of the CGI severity and improvement scales as measures of clinical effectiveness suitable for routine clinical use. J Eval Clin Pract. 2008 Dec;14(6):979-83. doi: 10.1111/j.1365-2753.2007.00921.x. Epub 2008 May 2. PMID 18462279
- [Background] de Looff P, Noordzij ML, Moerbeek M, Nijman H, Didden R, Embregts P. Changes in heart rate and skin conductance in the 30 min preceding aggressive behavior. Psychophysiology. 2019 Oct;56(10):e13420. doi: 10.1111/psyp.13420. Epub 2019 Jun 11. PMID 31184379
- [Background] Lifshitz M, Dwolatzky T, Press Y. Validation of the Hebrew version of the MoCA test as a screening instrument for the early detection of mild cognitive impairment in elderly individuals. J Geriatr Psychiatry Neurol. 2012 Sep;25(3):155-61. doi: 10.1177/0891988712457047. PMID 23124009
- [Background] Menghini L, Gianfranchi E, Cellini N, Patron E, Tagliabue M, Sarlo M. Stressing the accuracy: Wrist-worn wearable sensor validation over different conditions. Psychophysiology. 2019 Nov;56(11):e13441. doi: 10.1111/psyp.13441. Epub 2019 Jul 23. PMID 31332802
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Salzmann-Erikson M, Yifter L. Risk Factors and Triggers That May Result in Patient-Initiated Violence on Inpatient Psychiatric Units: An Integrative Review. Clin Nurs Res. 2020 Sep;29(7):504-520. doi: 10.1177/1054773818823333. Epub 2019 Jan 22. PMID 30666885
- [Background] Hedlund Lindberg M, Samuelsson M, Perseius KI, Bjorkdahl A. The experiences of patients in using sensory rooms in psychiatric inpatient care. Int J Ment Health Nurs. 2019 Aug;28(4):930-939. doi: 10.1111/inm.12593. Epub 2019 Mar 31. PMID 30931543
- [Background] Chalmers A, Harrison S, Mollison K, Molloy N, Gray K. Establishing sensory-based approaches in mental health inpatient care: a multidisciplinary approach. Australas Psychiatry. 2012 Feb;20(1):35-9. doi: 10.1177/1039856211430146. Epub 2012 Jan 5. PMID 22357673
- [Background] Wiglesworth S, Farnworth L. An Exploration of the Use of a Sensory Room in a Forensic Mental Health Setting: Staff and Patient Perspectives. Occup Ther Int. 2016 Sep;23(3):255-64. doi: 10.1002/oti.1428. Epub 2016 May 29. PMID 27237722
- See also: Skin conductance, heart rate and aggressive behavior type — http://doi.org/10.1016/j.biopsycho.2018.12.012
- See also: Sensory modulation disorder (SMD) and pain: a new perspective. — http://doi.org/10.3389/fnint.2019.00027
- See also: The effects of the use of the sensory room in psychiatry — http://www.ot-innovations.com/wp-ontent/uploads/2014/09/qi_study_sensory_room.pdf
- See also: The responsiveness of the Hamilton depression rating scale. — http://doi.org/10.1016/S0022-3956(99)00037-0
- See also: Predicting Depression and Anxiety Mood by Wrist-Worn Sleep Sensor — http://doi.org/10.1109/PerComWorkshops48775.2020.9156176
- See also: Autonomic nervous system activity in emotion: A review — http://doi.org/10.1016/j.biopsycho.2010.03.010
- See also: Linking the PANSS, BPRS, and CGI: clinical implications — http://doi.org/10.1038/sj.npp.1301147
- See also: Validation of the Empatica E4 wristband. — http://doi.org/10.1109/EMBSISC.2016.7508621
- See also: Pain sensitivity can be assessed by self-rating: Development and validation of the Pain Sensitivity Questionnaire — http://doi.org/10.1016/j.pain.2009.06.020
- See also: Validity of the Empatica E4 Wristband to Measure Heart Rate Variability (HRV) Parameters: A Comparison to Electrocardiography (ECG). — http://doi.org/10.1007/s10916-020-01648-w
- See also: Epidemiology of pain and relation to psychiatric disorders. — http://doi.org/10.1016/j.pnpbp.2017.05.012
- See also: Wearable devices and their applications in surgical robot control and p-medicine — http://doi.org/10.1109/CSCWD.2016.7566067
- See also: Sensory modulation and daily-life participation in people with schizophrenia. — http://doi.org/10.1016/j.comppsych.2014.12.009